CLINICAL TRIAL: NCT00198848
Title: Iron Supplementation Among Adolescent Girls in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H.32.04.11.22.A2; S3433-23/23 (ASPH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2006-01

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Adolescent girls; India
MeSH Terms: conditions — Anemia, Iron-Deficiency

INTERVENTIONS:
Drug: Iron-folic acid supplement

SUMMARY:
This study will implement and evaluate a community-based intervention to distribute and promote consumption of weekly iron-folic acid supplements and to provide nutrition education to reduce the prevalence of iron deficiency anemia among adolescent girls in West Bengal, India.

ELIGIBILITY:
Inclusion Criteria:

* Girl 12-19 years of age
* Resides in study area

Exclusion Criteria:

* Does not reside in study area

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2800 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia after 1 year of intervention

SECONDARY OUTCOMES:
Knowledge of anemia
Practices regarding treatment and prevention of anemia
Knowledge of iron supplements
Practices regarding iron supplements
Dietary iron intake

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Dreyfuss, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Child In Need Institute, Kolkata, West Bengal, India